CLINICAL TRIAL: NCT00831181
Title: A Phase II Open-labeled, Prospective Study to Determine the Efficacy of Preoperative Chemoradiation With Oxaliplatin/5-FU in Locally Advanced Rectal Cancer Followed by Total Mesorectal Excision and FOLFOX6
Brief Title: Neo-adjuvant Chemoradiation With Oxaliplatin/5-FU in Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000633360; BIMCP-OX-08-006 (Registry Identifier: BIMCP-OX-08-006); AVENTIS-BIMCP-OX-08-006 (Other Grant/Funding Number: AVENTIS-BIMCP-OX-08-006)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Results first posted 2018-03-20 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative Chemoradiation (Experimental): Preoperative Chemoradiation with oxaliplatin/5-FU followed by mesorectal excision and 5-FU / leucovorin (FOLFOX 6)
  Interventions: Drug: 5-FU; Drug: Oxaliplatin; Drug: leucovorin; Procedure: mesorectal excision

INTERVENTIONS:
Drug: 5-FU — 5-FU: continuous infusion via portable pump during all RT (approximately 33 days)
  Other Names: fluorouracil
Drug: Oxaliplatin — Oxaliplatin: 50mg/m2 weekly dosing during RT (Day 1)
  Other Names: Eloxatin
Drug: leucovorin — Folinic Acid (Leucovorin): 400 mg/m2; 2-hour IV infusion simultaneously with oxaliplatin
  Other Names: Folinic Acid
Procedure: mesorectal excision — mesorectal excision

SUMMARY:
RATIONALE: 5FU based neoadjuvant chemoradiation (nCRT) is the standard of care for Stage II/III rectal cancer. Pathologic complete response (pCR) and downstaging have been associated with improved outcomes. The addition of oxaliplatin (OXA) to neoadjuvant therapy may reduce distant disease recurrence. Adjuvant treatment with OXA for rectal cancer has been motivated by benefits demonstrated in stage III colon cancer.

Objective: To determine the feasibility, toxicity, and efficacy of preoperative OXA/5FU and RT followed by total mesorectal excision (TME) and adjuvant

PURPOSE: This phase II trial is studying the side effects and how well giving neo-adjuvant combination chemotherapy with radiation works in treating patients undergoing surgery for rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the complete pathologic response rate in patients with rectal cancer treated with radiation, modified neoadjuvant FOLFOX 6 chemotherapy followed by total mesorectal excision and adjuvant modified FOLFOX 6 chemotherapy.

Secondary

* To observe the overall pathologic response rate in these patients.
* To correlate pathologic staging with preoperative ultrasound and pelvic MRI staging.
* To assess toxic side effects of these regimens in these patients.
* To assess patterns of disease relapse, disease-free survival outcomes, and overall survival outcomes of these patients.

OUTLINE:

Patients with stage II/III rectal cancer were treated with OXA 60mg/m2 weekly continuous infusion 5FU of 225 mg/m2/d d1-5 with pelvic RT of 1.8Gy/d for 28 doses. Adjuvant therapy consisted of 6 cycles of biweekly FOLFOX6.

Surgery: Patients undergo total mesorectal excision by anterior resection or an abdominal perineal resection within 4 weeks after completion of neoadjuvant therapy.

Adjuvant therapy: Within 4 weeks after surgery, patients receive modified FOLFOX 6 chemotherapy comprising oxaliplatin and leucovorin calcium IV over 2 hours on day 1 and continuous fluorouracil IV over 46 hours on days 1-2. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality of life assessment questionnaires at baseline and at each follow-up visit.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria

* Histologically proven adenocarcinoma of the rectum with no distant metastases.
* T3-4N0M0, TanyN1-3M0 assessed by clinical exam, TRUS, MRI and CT
* The distal border of the tumor must be at or below the peritoneal reflection, defined as within 12 centimeters of the anal verge by protoscopic examination.
* No prior chemotherapy or pelvic irradiation.
* ECOG performance status 0-1
* Age 18 to 70 years
* ANC >= 1500/mm3 and platelets >= 100,000/mm3
* Serum creatinine <= 1.5 x ULN; bilirubin <= 1.5 x ULN; ALT<= 2.5 x ULN

Exclusion Criteria

* Pregnant or lactating females; patients not practicing active contraception while sexually active.
* No other serious medical condition
* A psychiatric disorder that would prohibit the subject from participating fully.
* Peripheral neuropathy > grade 1
* History within the past 5 years of a cancer diagnosis except for non-melanomatous skin cancers or in situ cervix carcinoma.
* HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kozuch, MD, Principal Investigator — Beth Israel Medical Center
Locations (2):
- United States (2):
  - Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York
  - St. Luke's-Roosevelt Hospital Center - Roosevelt Division, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 2004-2009 from the oncology practice at Beth Israel and Roosevelt Hospitals.
Groups:
- Oxaliplatin/5-FU Followed by Mesorectal Excision and FOLFOX 6: Preoperative Chemoradiation with oxaliplatin/5-FU followed by mesorectal excision and FOLFOX 6:
  Preoperative therapy: Oxaliplatin 60 mg/m2 weekly dosing during radiation with continuous infusion 5-FU 225 mg/m2/d Monday through Friday for a total of 96 hours per week each week of radiation (approximately 6-7 weeks). Radiation dose will be 50-54Gy with possible intraoperative (IORT) radiation (10-12Gy).
  Surgery: Total Mesorectal Excision
  Postoperative therapy: FOLFOX6 every 2 weeks for 6 cycles (3 months)
Period: Overall Study
Arm/Group | Oxaliplatin/5-FU Followed by Mesorectal Excision and FOLFOX 6
Started | 27
Completed | 15
Not Completed | 12
Not completed — Adverse Event | 12

BASELINE CHARACTERISTICS:
Groups:
- Chemoradiation,Surgery, Chemotherapy: Preoperative Chemoradiation with oxaliplatin/5-FU followed by mesorectal excision and FOLFOX 6
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response and Complete Response
Description: Pathologic Response and Complete Response to preoperative therapy will be determined at the time of surgical resection. All grossly visible areas of ulceration and/or induration with be measured and submitted for histological evaluation.
  The unit of measure is the tumor response rate to preoperative chemoradiation.
  Pathologic complete response (pCR) is defined as no evidence of invasive tumor cells on pathologic examination of the primary rectal cancer.
  Tumor regression grade (TRG) will be quantitated into five grades:
  TRG 1 (complete regression) -absence of residual cancer and fibrosis extending from the site of original tumor through the layers of the rectal wall.
  TRG 2 characterized by the presence of rare residual cancer cells scattered through the fibrosis.
  TRG 3 characterized by an increase in the number of residual cancer cells, but fibrosis still predominant.
  TRG 4 -residual cancer outgrowing fibrosis. TRG 5 characterized by absence of regressive changes.
Time Frame: Total mesorectal excision (TME) participants were evaluated at the time of surgical resection, an average of 3.5 months
Population: Number of subjects undergoing TME
Measure: Number; unit: Participants
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
Participants | 3

2. Secondary Outcome: Treatment Toxicity
Description: Toxicity was assessed weekly during neoadjuvant chemotherapy and radiation therapy, bi-weekly during adjuvant FOLFOX therapy.
Time Frame: Weekly during chemoradiation treatment (3 months). Bi-weekly during adjuvant FOLFOX therapy (3.5 months).
Population: According to the citation J Clin Oncol 28,2010 (suppl; abstract e14128): acute grade 3-4 toxicities occurred in 16 patients, mainly hypersensitivity reactions and OXA associated peripheral neuropathy.
Measure: Number; unit: patients
Groups:
- Chemoradiation,Surgery, Chemotherapy: Preoperative Chemoradiation with oxaliplatin/5-FU followed by mesorectal excision and FOLFOX 6:
  Preoperative therapy: Oxaliplatin 60 mg/m2 weekly dosing during radiation with continuous infusion 5-FU 225 mg/m2/d Monday through Friday for a total of 96 hours per week each week of radiation (approximately 6-7 weeks). Radiation dose will be 50-54Gy with possible intraoperative (IORT) radiation (10-12Gy).
  Surgery: Total Mesorectal Excision
  Postoperative therapy: FOLFOX6 every 2 weeks for 6 cycles (3 months)
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 27
patients | 16

3. Secondary Outcome: Complete Resectability Rates
Description: Complete resectability rates assessed by circumferential margin.
Time Frame: Total mesorectal excision (TME) participants were evaluated at the time of surgical resection, 3 months after beginning of chemoradiation treatment.
Population: Out of the 27 patients enrolled, a total 23 underwent TME.
Measure: Number; unit: patient
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
patient | 3

4. Secondary Outcome: Local Regional Control
Description: subjects were followed for median of 22 months post-surgery
Time Frame: median follow-up 22 months post-TME
Population: Out of the 27 patients enrolled, a total 23 underwent TME and were assessed for local regional control.
Measure: Number; unit: patient
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
patient | 21

5. Secondary Outcome: Disease-free Survival
Time Frame: median 22 months follow-up
Population: Out of the 27 patients enrolled, a total 23 underwent TME and were assessed for disease-free survival.
Measure: Number; unit: participants
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
participants | 16

6. Secondary Outcome: Overall Survival
Time Frame: median follow-up 22 months
Population: Patients who completed treatment
Measure: Number; unit: participants
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
participants | 21

7. Secondary Outcome: Patterns of Disease Failure, Including Local Recurrence and Distant Metastasis Assessed by CT Scan
Time Frame: median follow-up 22 months
Population: Out of the 27 patients enrolled, a total 23 underwent TME and were assessed for patterns of disease failure.
Measure: Number; unit: patients
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
patients | 2

8. Secondary Outcome: Number of Participants With Comparison of Preoperative Stage With Post-treatment Pathologic Stage
Description: Thin-section high resolution pelvic MRI was used to image the tumor prior to chemoradiation and repeated prior to surgery, and then compared to post-treatment pathological stage.
Time Frame: as for outcome 3
Population: Out of the 27 patients enrolled, a total 23 underwent TME. These 23 patients were included for comparison of preoperative stage and post-treatment pathologic stage.
Measure: Number; unit: patient
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Number analyzed (Participants) | 23
patient | 13

ADVERSE EVENTS:
Arm/Group | Chemoradiation,Surgery, Chemotherapy
Serious Adverse Events (participants affected / at risk) | 16/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemoradiation,Surgery, Chemotherapy (N=27)
peripheral neuropathy (Nervous system disorders) | 10 (10)
oxaliplatin intolerance (Immune system disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes